CLINICAL TRIAL: NCT00703664
Title: Phase II Trial of Bortezomib and Vorinostat in Mantle Cell and Diffuse Large B-Cell Lymphomas
Brief Title: Bortezomib and Vorinostat in Treating Patients With Recurrent Mantle Cell Lymphoma or Recurrent and/or Refractory Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00275; NCI-2009-00275 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000598308; MCC-15428 (Other: Moffitt Cancer Center); 8064 (Other: CTEP); N01CM00071 (NIH); N01CM00100 (NIH); N01CM62201 (NIH); N01CM62204 (NIH); N01CM62208 (NIH); P30CA076292 (NIH)
Record Dates: First submitted 2008-06-20; First posted 2008-06-23 (Estimated); Results first posted 2018-08-07 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-07

CONDITIONS: Recurrent Mantle Cell Lymphoma; Recurrent Non-Hodgkin Lymphoma
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Lymphoma, Non-Hodgkin | interventions — Bortezomib; Vorinostat

ARMS (1):
- Treatment (vorinostat, bortezomib) (Experimental): Participants receive vorinostat orally (PO) once daily (QD) on days 1-5 and 8-12. Participants also receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Vorinostat precedes bortezomib on days of concurrent administration. Courses repeat every 3 weeks in the absence of disease progression - or unacceptable toxicity. After completion of study therapy, participants are followed periodically.
  Treatment arm consists of 3 cohorts, all receiving the same treatment:
  A: Mantle Cell Lymphoma (MCL) - with no prior bortezomib.
  B: Mantle Cell Lymphoma (MCL) - with no prior bortezomib.
  C: Diffuse Large B-Cell Lymphoma (DLBCL) - with no prior bortezomib.
  Interventions: Drug: Bortezomib; Other: Laboratory Biomarker Analysis; Drug: Vorinostat

INTERVENTIONS:
Drug: Bortezomib — Bortezomib: 1.3 mg/m^2/d IV days 1, 4, 8, and 11.
  Other Names: [(1R)-3-Methyl-1-[[(2S)-1-oxo-3-phenyl-2-[(pyrazinylcarbonyl)amino]propyl]amino]butyl]boronic Acid; LDP 341; MLN341; PS-341; PS341; Velcade
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Vorinostat — Vorinostat: 400 mg (total daily dose as a single dose) days 1-5 and 8-12.
  Other Names: L-001079038; MSK-390; SAHA; Suberanilohydroxamic Acid; Suberoylanilide Hydroxamic Acid; Zolinza

SUMMARY:
This phase II trial studies how well bortezomib and vorinostat work in treating patients with recurrent mantle cell lymphoma or recurrent and/or refractory diffuse large B-cell lymphoma. Bortezomib and vorinostat may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
This was a multicenter, non-randomized phase 2 trial using a Simon two-stage design with 3 cohorts.

PRIMARY OBJECTIVES:

I. Estimate the response rates of mantle cell and diffuse large B-cell lymphomas to bortezomib and vorinostat combination therapy.

SECONDARY OBJECTIVES:

I. Assess the safety and tolerability of the study regimen. II. Observe progression-free survival and response durations. III. Observe the relationship between pretreatment lymphoma cell nuclear v-rel reticuloendotheliosis viral oncogene homolog A (relA) and response.

OUTLINE:

Patients receive vorinostat orally (PO) once daily (QD) on days 1-5 and 8-12. Patients also receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed mantle cell or diffuse large B-cell lymphoma; histological material must be available for central pathological review; unstained histological material -- slides or blocks -- must be available for correlative studies; archived material from previous biopsies is acceptable, unless a patient's lymphoma has been known to undergo histological transformation in the past, in which case a repeat biopsy to confirm histology prior to enrollment is required; availability of material must be confirmed at the time of registration, but material may be submitted subsequent to registration and initiation of study treatment
* Measurable disease according to the Revised Response Criteria for Malignant Lymphoma; this requires at least one lesion greater than 1.0 cm in diameter in both the long and short axis as measured by spiral computed tomography (CT) scan or physical exam
* Prior allogeneic stem cell transplant is allowed provided that all of the following conditions are met:

  * >= 6 months have elapsed since allogeneic transplant
  * No graft vs. host disease (GVHD) is present
  * Not currently on immunosuppressive therapy
* Prior therapy:

  * Mantle cell lymphoma:

    * Previously treated or untreated
    * No prior bortezomib
  * Diffuse large B-cell lymphoma:

    * At least one prior systemic therapy
    * No prior bortezomib

      * Note: Not intended for patients in first relapse who are candidates for high dose therapy with stem cell support
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2
* Able to tolerate loperamide or other anti-diarrheal medications
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 75 x 10^9/L
* Total bilirubin =< 1.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transferase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x institutional upper limit of normal
* Creatinine within normal institutional limits or calculated creatinine clearance >= 60 mL/min according to the Cockcroft-Gault formula
* For patients with known human immunodeficiency virus (HIV) infection, a cluster of differentiation (CD)4 count >= 0.5 x 10^9/L
* For patients whose last treatment included bendamustine or fludarabine, a CD4 count >= 0.4 x 10^9/L
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation and to report pregnancy or suspected pregnancy while participating in the study
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Chemotherapy or large field radiotherapy within 3 weeks prior to entering the study
* Prior histone deacetylase inhibitor as cancer treatment
* Concurrent treatment with other investigational agents
* Plans for other concurrent cancer treatment; if steroids for cancer control have been used, patients must be off these agents for >= 1 week before starting treatment; exception: maintenance therapy for non-malignant disease with prednisone or steroid equivalent dose < 10 mg/day is permitted
* History of brain metastasis including leptomeningeal metastasis
* Grade >= 2 neuropathy, regardless of cause
* Unable to take oral medications
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to bortezomib or vorinostat
* Not sufficiently recovered from previous treatment
* Medical or other condition (for example: uncontrolled infection; potentially life threatening changes on electrocardiogram [EKG]) or concurrent treatment (for example, marrow suppressive agents such as zidovudine) that represents an inappropriate risk to the patient or likely would compromise achievement of the primary study objective; patients should be closely monitored when given bortezomib in combination with the cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors and inducers
* Pregnant women are excluded from this study; breastfeeding should be discontinued
* Active concurrent malignancy, except adequately treated non-melanoma skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2008-07-09 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2017-12-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Beata Holkova, Principal Investigator — Massey Cancer Center
Locations (12):
- United States (12):
  - Moffitt Cancer Center, Tampa, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - University of Maryland/Greenebaum Cancer Center, Baltimore, Maryland
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Weill Medical College of Cornell University, New York, New York
  - Montefiore Medical Center-Weiler Hospital, The Bronx, New York
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Virginia Commonwealth University/Massey Cancer Center, Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 participating cancer center sites in the United States, from July 2008 through December 2013.
Groups:
- Treatment: Cohort A - MCL; No Prior Bortezomib: Mantle Cell Lymphoma (MCL): Treatment (vorinostat, bortezomib). Participants receive vorinostat orally (PO) once daily (QD) on days 1-5 and 8-12. Participants also receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Vorinostat precedes bortezomib on days of concurrent administration. Courses repeat every 3 weeks in the absence of disease progression - or unacceptable toxicity. After completion of study therapy, participants are followed periodically.
- Treatment: Cohort B - MCL; Prior Bortezomib: Mantle Cell Lymphoma MCL: Treatment (vorinostat, bortezomib). Participants receive vorinostat orally (PO) once daily (QD) on days 1-5 and 8-12. Participants also receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Vorinostat precedes bortezomib on days of concurrent administration. Courses repeat every 3 weeks in the absence of disease progression - or unacceptable toxicity. After completion of study therapy, participants are followed periodically.
- Treatment: Cohort C - DLBCL; No Prior Bortezomib: Diffuse Large B-Cell Lymphoma (DLBCL): Treatment (vorinostat, bortezomib). Participants receive vorinostat orally (PO) once daily (QD) on days 1-5 and 8-12. Participants also receive bortezomib intravenously (IV) over 3-5 seconds on days 1, 4, 8, and 11. Vorinostat precedes bortezomib on days of concurrent administration. Courses repeat every 3 weeks in the absence of disease progression - or unacceptable toxicity. After completion of study therapy, participants are followed periodically.
Period: Overall Study
Arm/Group | Treatment: Cohort A - MCL; No Prior Bortezomib | Treatment: Cohort B - MCL; Prior Bortezomib | Treatment: Cohort C - DLBCL; No Prior Bortezomib
Started | 22 | 4 | 39
Completed | 22 | 4 | 39
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who received treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment: Cohort A - MCL; No Prior Bortezomib | Treatment: Cohort B - MCL; Prior Bortezomib | Treatment: Cohort C - DLBCL; No Prior Bortezomib | Total
Number analyzed (Participants) | 22 | 4 | 39 | 65
Age, Continuous [Median (Full Range); unit: years] | 64 [48 to 72] | 63 [58 to 78] | 57 [29 to 89] | 60 [29 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 0 | 13 | 18
  Male | 17 | 4 | 26 | 47
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 5 | 7
  White | 19 | 4 | 30 | 53
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 4 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 22 | 4 | 39 | 65
Eastern Cooperative Oncology Group (ECOG) Status [Count of Participants; unit: Participants] — ECOG Status 0: Normal activity. Fully active, able to carry on all pre-disease performance without restriction. ECOG Status 1: Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (e.g., light housework, office work). ECOG Status 2: In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    Status: 0 | 13 | 3 | 11 | 27
    Status: 1 | 9 | 1 | 19 | 29
    Status: 2 | 0 | 0 | 9 | 9

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR: Complete Response (CR) + Partial Response (PR) assessed according to the Revised Response Criteria for Malignant Lymphoma.
Time Frame: Up to 9 years
Population: All participants.
Measure: Number; unit: percentage of participants
Groups:
- Cohort A - MCL: Mantle Cell Lymphoma (MCL): Treatment (vorinostat, bortezomib).
- Cohort B - MCL: Mantle Cell Lymphoma MCL: Treatment (vorinostat, bortezomib).
- Cohort C - DLBCL: Diffuse Large B-Cell Lymphoma (DLBCL): Treatment (vorinostat, bortezomib).
Arm/Group | Cohort A - MCL | Cohort B - MCL | Cohort C - DLBCL
Number analyzed (Participants) | 22 | 4 | 39
percentage of participants | 31.8 | 0 | 7.7

2. Secondary Outcome: Best Response
Description: Number of participants per category: Partial Response (PR), Stable Disease (SD), Progressive Disease (PD). PR: Regression of measurable disease and no new sites. SD: Failure to attain Complete Response (CR), /PR or PD. Relapsed or Progressive Disease: Any new lesion or increase by ≥ 50% of previously involved sites from nadir.
Time Frame: Up to 9 years
Population: All participants evaluable and available at time of assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort A - MCL | Cohort B - MCL | Cohort C - DLBCL
Number analyzed (Participants) | 19 | 4 | 34
Participants
  Partial Response | 7 | 0 | 3
  Stable Disease | 5 | 2 | 8
  Progressive Disease | 7 | 2 | 23

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Median progression-free survival in months per cohort.
Time Frame: Up to 9 years
Population: All evaluable participants at time of analysis. Cohort B was closed early due to lack of accrual.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort A - MCL | Cohort B - MCL | Cohort C - DLBCL
Number analyzed (Participants) | 22 | 0 | 39
months | 7.6 [2.2 to NA] — not reached |  | 1.8 [1.4 to 2.3]

4. Secondary Outcome: Duration of Partial Response
Description: Median duration of response per cohort.
Time Frame: Up to 9 years
Population: All participants with Partial Response.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A - MCL | Cohort B - MCL | Cohort C - DLBCL
Number analyzed (Participants) | 7 | 0 | 3
months | 4.2 [0.13 to 16.9] |  | 2.1 [1.34 to 2.13]

5. Secondary Outcome: Duration of Stable Disease
Description: Median duration of stable disease per cohort.
Time Frame: Up to 9 years
Population: All participants with stable disease.
Measure: Median (Full Range); unit: months
Arm/Group | Cohort A - MCL | Cohort B - MCL | Cohort C - DLBCL
Number analyzed (Participants) | 5 | 2 | 8
months | 3.8 [0.3 to 13.4] | 3.8 [3.5 to 4] | 1.3 [0.03 to 6.97]

ADVERSE EVENTS:
Time Frame: 5 years
Description: NCI Common Terminology Criteria for Adverse Events (CTCAE) v3.0 was used for reporting adverse events until April 1, 2011, when mandatory conversion to CTCAE v4.0 supervened. Response was assessed using the Revised Response Criteria for Malignant Lymphoma.
Arm/Group | Cohort A - MCL | Cohort B - MCL | Cohort C - DLBCL
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/4 | 4/39
Serious Adverse Events (participants affected / at risk) | 9/22 | 1/4 | 22/39
Other Adverse Events (participants affected / at risk) | 22/22 | 4/4 | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - MCL (N=22) | Cohort B - MCL (N=4) | Cohort C - DLBCL (N=39)
Multi-organ failure - Death (General disorders) | 0 (0) | 0 (0) | 1 (1) — Possibly related to bortezomib, vorinostat, or progression of DLBCL.
Neoplasms benign, malignant and unspecified - Death (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Unlikely to be related to study drug treatment.
Multi-organ failure (General disorders) | 0 (0) | 0 (0) | 1 (1) — Unrelated to study treatment.
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Ventricular arrhythmia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Dry Eye (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eye disorders - Other, Chalazion (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders - Other, Cramping (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Chills (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema limbs (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1)
Fever (General disorders) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infectionsand infestations - Other (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Creatinine increased (Investigations) | 1 (1) | 0 (0) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1) | 1 (2)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Platelet count decreased (Investigations) | 0 (0) | 0 (0) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 3 (3)
Hypercalcemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (3)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 1 (2)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Nervous system disorders - Other (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 6 (6)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 0 (0) | 3 (3)
Thromboembolic event (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort A - MCL (N=22) | Cohort B - MCL (N=4) | Cohort C - DLBCL (N=39)
Diarrhea (Gastrointestinal disorders) | 20 (54) | 2 (2) | 24 (46)
Nausea (Gastrointestinal disorders) | 14 (33) | 2 (2) | 20 (47)
Vomiting (Gastrointestinal disorders) | 10 (16) | 0 (0) | 14 (24)
Constipation (Gastrointestinal disorders) | 7 (8) | 1 (1) | 12 (15)
Abdominal pain (Gastrointestinal disorders) | 5 (6) | 1 (1) | 10 (12)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 5 (5)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (2)
Abdominal distension (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastroparesis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Platelet count decreased (Investigations) | 18 (126) | 3 (5) | 26 (141)
Lymphocyte count decreased (Investigations) | 11 (30) | 1 (1) | 20 (65)
White blood cell decreased (Investigations) | 13 (32) | 1 (1) | 14 (65)
Neutrophil count decreased (Investigations) | 10 (19) | 0 (0) | 12 (32)
Creatinine increased (Investigations) | 7 (19) | 1 (3) | 12 (42)
Aspartate aminotransferase increased (Investigations) | 3 (6) | 0 (0) | 7 (10)
Alanine aminotransferase increased (Investigations) | 3 (5) | 0 (0) | 5 (9)
Alkaline phosphatase increased (Investigations) | 0 (0) | 0 (0) | 6 (8)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1) | 0 (0) | 1 (1)
Weight loss (Investigations) | 3 (3) | 0 (0) | 1 (1)
Investigations - Other, specify (Investigations) | 1 (1) | 0 (0) | 2 (6)
INR increased (Investigations) | 0 (0) | 1 (1) | 1 (1)
Weight gain (Investigations) | 0 (0) | 1 (1) | 1 (1)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Cardiac troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (3)
Cholesterol high (Investigations) | 0 (0) | 0 (0) | 1 (1)
CPK increased (Investigations) | 0 (0) | 0 (0) | 1 (2)
Anorexia (Metabolism and nutrition disorders) | 11 (11) | 0 (0) | 15 (23)
Hyperglycemia (Metabolism and nutrition disorders) | 5 (7) | 3 (6) | 14 (25)
Hyponatremia (Metabolism and nutrition disorders) | 5 (14) | 0 (0) | 11 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 5 (11) | 0 (0) | 10 (17)
Dehydration (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 4 (4)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) | 9 (12)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5) | 0 (0) | 6 (17)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (4) | 0 (0) | 6 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 6 (9)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 3 (4)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0) | 1 (1)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0) | 3 (4)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (4)
Hyperuricemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 2 (2)
Fatigue (General disorders) | 18 (39) | 1 (4) | 22 (48)
Chills (General disorders) | 7 (10) | 0 (0) | 2 (3)
Edema limbs (General disorders) | 2 (2) | 0 (0) | 5 (6)
Fever (General disorders) | 2 (3) | 0 (0) | 6 (9)
Pain (General disorders) | 2 (2) | 0 (0) | 6 (7)
Malaise (General disorders) | 2 (3) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Edema trunk (General disorders) | 0 (0) | 0 (0) | 1 (1)
Facial pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Irritability (General disorders) | 0 (0) | 1 (1) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 10 (20) | 1 (2) | 10 (12)
Dizziness (Nervous system disorders) | 12 (16) | 1 (1) | 7 (7)
Headache (Nervous system disorders) | 2 (2) | 1 (1) | 11 (15)
Dysgeusia (Nervous system disorders) | 3 (3) | 0 (0) | 1 (2)
Paresthesia (Nervous system disorders) | 2 (2) | 0 (0) | 2 (2)
Peripheral motor neuropathy (Nervous system disorders) | 1 (2) | 0 (0) | 2 (2)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (3) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 7 (26) | 1 (1) | 20 (70)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (1)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (8) | 0 (0) | 3 (6)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (4) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 (6) | 0 (0) | 12 (15)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 2 (2) | 7 (8)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 2 (2)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (2)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 4 (4)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1) | 2 (2)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (3) | 0 (0) | 3 (3)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Periorbital edema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Scalp pain (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Skin induration (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Infections and infestations - Other, specify (Infections and infestations) | 2 (2) | 0 (0) | 1 (1)
Papulopustular rash (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (3) | 0 (0) | 1 (1)
Hepatitis viral (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Mucosal infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 4 (5) | 0 (0) | 5 (6)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0) | 3 (3)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 3 (4)
Agitation (Psychiatric disorders) | 0 (0) | 1 (2) | 1 (1)
Restlessness (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 3 (7) | 0 (0) | 4 (4)
Hypertension (Vascular disorders) | 2 (4) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0) | 1 (3)
Lymphedema (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Proteinuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1)
Urinary frequency (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 2 (2)
Urinary tract pain (Renal and urinary disorders) | 0 | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 3 (4)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Blurred vision (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Injury, poisoning and procedural complications - Other, specify (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune disorder (Immune system disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder fistula (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Cohort C met the 1st-stage efficacy endpoint to proceed to the 2nd stage but was closed with evidence that the 2nd-stage efficacy endpoint could not be achieved.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-04-10): https://cdn.clinicaltrials.gov/large-docs/64/NCT00703664/Prot_SAP_000.pdf